CLINICAL TRIAL: NCT00331175
Title: A Phase 1, Randomized, Placebo- And Positive Controlled Study To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Escalating Doses Of Intravenous Peptide YY3-36 In Otherwise Healthy Overweight Adult Subjects
Brief Title: Safety, Toleration and Pharmacokinetics of Single Intravenous Doses of Peptide YY in Overweight Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A9001292
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — peptide YY (3-36)

INTERVENTIONS:
Drug: Peptide YY3-36

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of single escalating doses of Peptide YY3-36 and to determine effects on food intake and serum hormones when administered by intravenous infusion to otherwise healthy overweight adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-35 kg/m2

Exclusion Criteria:

* Women of childbearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31
Dates: Start 2006-07; Study Completion 2006-12

PRIMARY OUTCOMES:
Food intake

SECONDARY OUTCOMES:
Plasma biomarkers, safety, toleration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001292&StudyName=Safety%2C+toleration+and+pharmacokinetics+of+single+intravenous+doses+of+Peptide+YY+in+overweight+adults